CLINICAL TRIAL: NCT06643169
Title: The Effect of Home Based Fall Prevention Program on Fall Rate Among Older Adults at High Risk of Falling
Brief Title: The Effect of Home Based Fall Prevention Program on Older Adults at High Risk of Falling
Acronym: HoBFaPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Feyza Demir Bozkurt, M.sC., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IUC-NURSE-FDB-01
Record Dates: First submitted 2024-10-13; First posted 2024-10-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Fall Prevention; Elderly; Home Based Care; Fall Risk
Keywords: high fall risk; elderly; fall prevention; home based

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): 8-week home-based fall prevention program with multifactorial intervention
  Interventions: Behavioral: home-based fall prevention program with multifactorial
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: home-based fall prevention program with multifactorial — * Health Education
  * Otago Exercises
  * Assessing and Organizing the Safe Home Environment
  Arms: Experimental Group

SUMMARY:
Fall prevention programs that implement and evaluate fall rates, balance status, accidents related to falls and hospital admissions, exercise status, muscle strength, fear of falling, and quality of life can be effective interventions for healthy aging by minimizing the risk of falls in elderly individuals. In this doctoral dissertation study, it was aimed to evaluate the effect of a nurse-led home-based fall prevention program on fall rate, balance level, fall risk score, fear of falling, number of hospital admissions due to falls, quality of life, and in-home safety conditions in older adults with high fall risk.

DETAILED DESCRIPTION:
Falls are a significant public health problem frequently seen among older people. Approximately one-third of individuals aged 65 years and older fall every year, and fall-related deaths are the leading cause of death in the elderly. According to World Health Organization (WHO) data, between 28% and 35% of adults over 65 fall every year; this rate increases to 42% from age 70. Falls and complications arising from falls are an essential problem for nurses working in primary care. In many countries, primary care nurses play an active role in meeting the health needs of the aging population. However, nurses are the health professionals who spend the most time with individuals, especially elderly individuals, who come to receive health services in primary healthcare organizations.

Nurses can assess the fall risk of elderly individuals with reliable screening tools at specific intervals. As a result, they can develop individualized nursing care plans by identifying existing and potential fall risks. Fall risk assessment in primary care and fall risk reduction practices planned after the assessment should be part of both the first health visit and subsequent visits. In the literature, nurse-led fall prevention programs are reported to be effective and promising for preventing falls for older individuals. In the future, nurses will have a more critical role in addressing older individuals' health problems and challenges. Nurses conduct much research involving evidence-based interventions to protect and promote health and manage diseases in various healthcare settings. Nursing science will continue to build the scientific evidence base for better clinical care and improved quality of life for the aging population. Specialist public health nurses also conduct various fall prevention programs for the elderly. It is reported that fall prevention programs reduce the fall rates and fear of falling, improve balance levels, increase quality of life, and positively affect the ability to maintain activities of daily living and live independently. Fall prevention programs that implement and evaluate fall rates, balance status, accident and hospital admissions related to falls, exercise status, muscle strength, fear of falling, and quality of life interventions in fall prevention programs can be an effective intervention for healthy aging by minimizing the risk of falls in elderly individuals. In this doctoral dissertation study, it was aimed to evaluate the effect of a nurse-led home-based fall prevention program on fall rate, balance level, fall risk score, fear of falling, number of hospital admissions due to falls, quality of life, and in-home safety conditions in older adults with high fall risk.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years and over with a high risk of falling (Those who score four and above on the Falls Risk Self-Assessment Scale will be determined as having a high risk of falling).
* To be examined by a physical therapist and to obtain consent that there is no harm in exercising (They will be referred to Bartın State Hospital and evaluated by a physical therapy specialist physician),
* Without a diagnosis of orthostatic hypotension,
* Elderly individuals who volunteered to participate in the study were identified.

Exclusion Criteria:

* Cardiovascular surgery in the last one year
* Diagnosis of orthostatic hypotension
* Having a neurological or neurodegenerative disease (such as Parkinson's dementia)
* Older people who exercise regularly,

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of falls | baseline, 2 months and 3 months
  elderly self-report with falls diary

SECONDARY OUTCOMES:
Balance level | baseline, 2 months and 3 months
  Berg Balance Scale:
  It consists of 14 items and each section is graded from 0 (bad) to 4 (best), measuring the level of dependency and/or independence during positions such as standing up from sitting, standing with feet together, standing in a full balance position, balancing on one leg, and the ability of the person to change position. A high score from the BBS indicates good balance. According to the scores obtained from this test, cases are divided into "high risk of falling, balance disorder (0-20 points)", "moderate risk of falling, acceptable balance (21-40 points)", "low risk of falling, good balance (41-56 points)".
Fall risk score | baseline, 2 months and 3 months
  Timed Up and Go Test: It is used to assess the risk of falling and mobility in the elderly. The TUG test is a balance test frequently used to assess functional mobility in frail elderly (70-84 years of age) living in the community. It was developed by Podsiadlo and Richardson in 1991. The test measures the speed during many functional maneuvers such as standing up, walking, turning and sitting down. In the test, the person is asked to stand up from the chair, walk 3 meters (10ft) at a safe and normal speed, turn around, walk back and sit down on the chair and the time is recorded in seconds. A shorter time indicates better balance and mobility skills. The starting position of the test should be standardized. In this study, it will be performed twice and the average will be taken. TUG is a simple, sensitive and specific test used to measure the probability of falling in the elderly.
Fear of falling | baseline, 2 months and 3 months
  International Falls Efficacy Scale (FES-I): Each item of the sixteen-item scale is rated between 1 and 4 points (I am not worried at all: 1 point, I am a little worried: 2 points, I am quite worried: 3 points, I am very worried: 4 points). The total scale score varies between 16 and 64, and a higher score indicates an increased fear of falling. FES-I is a scale that evaluates how much older individuals trust themselves in their daily living activities and shows their level of fear of falling.
Home environment assessment | baseline, 2 months and 3 months
  Fall-Related Home Safety Conditions Assessment Form: Developed by Belgin and Lok in 2012, the form evaluates the features that may pose a risk for elderly individuals to fall inside the home. The form consists of a total of 41 questions and their distribution to the areas is as follows; living room 7, kitchen 6, bedroom 7, bathroom/toilet 9, stairs 10 and corridor 4 questions. Each question is scored as Yes "0", No "1" and GY (no observation) "0" if the area planned to be observed is not inside the house, according to the risk in the examined area. The highest score received from the form is "41" and the lowest is "0". High scores indicate a high risk of falling, and a "0" score means no risk.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Secginli, Prof.Dr., Study Director — selda.secginli@atlas.edu.tr
Locations (1):
- Primary Health Center, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No